CLINICAL TRIAL: NCT03119454
Title: Evaluation of Pharmacokinetic Parameters of "Diprospan"
Brief Title: "Corticoid-16" in Long Term When Administered Systemically in Patients in Routine Medical Practice
Status: Completed | Type: Observational
Sponsor: Federal State Budgetary Scientific Institution, Scientific Research Institute of Rheumatology (Other)
Collaborators: Institute of Biomedical Chemistry, Russia (Other); The League of Clinical Research, Russia (Other)
Responsible Party: Sponsor
Other Study IDs: RU-FANO-10-16
Record Dates: First submitted 2016-12-09; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2016-12

CONDITIONS: Pharmacological Action
MeSH Terms: interventions — betamethasone dipropionate, betamethasone sodium phosphate drug combination; Betamethasone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients receiving diprospan: Patients who are receiving diprospan in standard therapy of their existing disease, or multiple times, but following the introduction of diprospan is planned no earlier than 28 days after the first administration.
  Interventions: Drug: Diprospan
- Control subjects: Patients or healthy volunteers who had not received systemic or local corticosteroids in the last 12 weeks before the screening visit.

INTERVENTIONS:
Drug: Diprospan — Intramuscular
  Other Names: Betamethasone
  Groups: Patients receiving diprospan

SUMMARY:
Evaluation of pharmacokinetic parameters of diprospan in long term when administered systemically in patients in routine medical practice.

Applied research project.

Design: open-comparative prospective cohort study.

Two groups of subjects:

* patients who are receiving diprospan in standard therapy of their existing disease, or multiple times, but following the introduction of diprospan is planned no earlier than 28 days after the first,
* control group of subjects for the study of pharmacokinetic parameters diprospan and its metabolites.

Objectives of the study: to evaluate the pharmacokinetic parameters of Diprospan in the long term when administered systemically in patients in routine practice.

DETAILED DESCRIPTION:
Design: Open-comparative prospective cohort study.

The study population: two groups of subjects

* first group: patients who are receiving diprospan in standard therapy of their existing disease, or multiple times, but following the introduction of diprospan is planned no earlier than 28 days after the first administration.
* second group: the control group of subjects for the study of pharmacokinetic parameters diprospan and its metabolites.

Intramuscular injection diprospan (suspension for injection) at a dose of 1 ml (7 mg) once.

Main objective of the study: to evaluate pharmacokinetic parameters of Diprospan in the long term when administered systemically in patients in routine practice.

Objectives of the study:

* to develop laboratory analytical method of quantifying the investigated substance (betamethasone) in human urine sensitive, selective and precise method using high performance liquid chromatography with tandem mass selective detection,
* analysis of quantitative content, evaluation of pharmacokinetic parameters of diprospan in the bioassay in patients with systemic intramuscular application in routine clinical practice in the Russian Federation,
* analysis of clinical patient data and pharmacokinetic parameters of study drug in the urine of patients,
* determination of minimum number of arbitration bioassay to store,
* preparation of recommendations for systemic use of glucocorticoids in athletes, in accordance with the requirements of the all-Russian anti-doping rules and the requirements of the anti-doping rules, approved by the international anti-doping authorities.

First group (patients receiving diprospan).

Stage 1: selection of study participants from a number of patients who are administered with Diprospan" at a dose of 1 ml (7 mg) intramuscularly as standard therapy of existing disease, or multiple times, but following introduction of "Diprospan" drug is planned no earlier than 28 days after the first.

Step 2: draw the original samples for pharmacokinetic studies, a single injection of the study medication as part of routine care.

Stage 3: Sampling in dynamics for pharmacokinetic studies; assessment of clinical and laboratory parameters after a single administration of the study drug.

Stage 4: evaluation of clinical examination data and pharmacokinetic study.

Second group (control).

Stage 1: selection of study participants from a number of patients or healthy volunteers who had not received systemic or local corticosteroids in the last 12 weeks before the screening visit.

Stage 2: drawing of samples for pharmacokinetic studies.

Primary endpoints:

• betamethasone concentration in urine.

Secondary endpoints:

* evaluation of articular status,
* overall assessment of the health status of the patient,
* overall assessment of disease activity, physician assessment of disease activity criteria for SDAI, CDAI, DAS-28.

Number of patients.

First group (the study of the pharmacokinetics of the drug "Diprrospan"): at least 20 patients (10 men and 10 women).

The second group (control): at least 20 patients (10 men and 10 women).

Safety monitoring In accordance with the order of the Health Ministry of Russia №757n "Approval of the Procedure for monitoring the safety of medicinal products for medical use, registration of adverse events, serious adverse reactions, unexpected adverse reactions in the use of drugs for medical use."

ELIGIBILITY:
Inclusion Criteria:

* Signed a voluntary informed consent form,
* Patients of both sexes aged 18 to 35 years old Caucasian,
* Verified diagnosis of rheumatoid arthritis according to criteria ACR \ EULAR 2010 or ankylosing spondylitis (axial spondyloarthritis) ASAS criteria for 2009 based on the data a detailed medical history, a standard clinical, laboratory and instrumental methods of examination,
* The presence of signs of active inflammation according to standard valuation techniques (for rheumatoid arthritis or DAS28 ≥3.2 CDAI≥10; for ankylosing spondylitis or BASDAI≥2.0 ASDAS≥1.3),
* If the patient gets authorized for use in the study antirheumatic drugs (except glucocorticoids other) for treatment of the underlying disease, they should be applied in stable doses for at least six weeks before the screening visit.
* BMI should be in the range of 18.0 to 30.0 kg / m 2 ,
* Consent to use adequate methods of contraception to patients during the study period.

Exclusion Criteria:

* Allergic history,
* Drug intolerance, hypersensitivity to any of the components "Diprospan" drug,
* Severe chronic cardiovascular, bronchopulmonary, endocrine and nervous systems (including mental) and diseases of the gastrointestinal tract (GIT), liver, kidney, blood, surgical procedures on the gastrointestinal tract (except appendectomy)
* Acute infectious, non-infectious and allergic diseases in less than 4 weeks prior to visit 1,
* A positive blood test for HIV, syphilis, hepatitis B and C,
* Systolic blood pressure measured at rest after 5 minutes of exposure in the "sitting" position, below 100 mm Hg. or above 140 mm Hg and / or diastolic blood pressure below 60 mm Hg or above 90 mm Hg,
* Heart rate below 40 beats / min,
* Hemoglobin <90 g / l (9 g / dl), or hematocrit less than 30%,
* White blood cells <3.0 x 10 9 / L,
* Absolute neutrophil count (ANC) <1.0 x 10 / L,
* Serum creatinine more than 0.132 mmol / L,
* Increased ALT and / or AST 1.5 upper limit of normal,
* Clinically significant (in the opinion of the investigator) ECG changes,
* The use of systemic or local corticosteroids for the treatment of the underlying disease for the last 12 weeks before the screening visit,
* Taking any medications, in addition to permissible under study
* Plasmapheresis in less than 14 days prior to study entry,
* Participation in a clinical trial of an unregistered in the Russian Federation of a drug or device for less than 3 months prior to the study,
* The inability or unwillingness of the patient to comply with the conditions of the study program,
* Any reason for that, according to the researcher, will prevent the participation of the patient in the study,
* Pregnant or lactating women (all women should have a negative pregnancy test on the day of screening).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients of both sexes aged 18 to 35 years old Caucasian,
  * verified diagnosis of rheumatoid arthritis according to criteria ACR \ EULAR 2010 or ankylosing spondylitis (axial spondyloarthritis) ASAS criteria for 2009 based on the data a detailed medical history, a standard clinical, laboratory and instrumental methods of examination.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-10; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Betamethasone concentration in urine | Day 28
  Quantitative determination of study drug (betamethasone) in human urine should be conducted sensitive, selective and precise method using high performance liquid chromatography with tandem mass selective detection (HPLC-MS / MS) with a detection mode permits fragment ions not more R <70K. laboratory analytical method should be developed for the measurement of betamethasone with the definition of the limit of not less than 7.5 ng / mL.

SECONDARY OUTCOMES:
Articular status (swelling) | Day 28
  Number of swollen joints
Articular status (pain) | Day 28
  Number of painful joints
Physician's assessment of disease activity | Day 28
  Visual analogue scale, mm
Simple disease activity index SDAI | Day 28
  Scale: remission; low activity; moderate activity; high activity
Clinical disease activity index CDAI | Day 28
  Scale: remission; low activity; moderate activity; high activity
Disease activity score DAS28 | Day 28
  Scale: remission; low activity; moderate activity; high activity

OTHER OUTCOMES:
Overall assessment of the health status of the patient by physician | Day 28
  Vital signs, physical examination, new diagnoses
Overall assessment of the health status of the patient by patient | Day 28
  Visual analogue scale, mm

REFERENCES:
- [Derived] Kopylov AT, Novikov AA, Kaysheva AL, Vykhodets IT, Karateev DE, Zgoda VG, Lisitsa AV. Quantitative assessment of betamethasone dual-acting formulation in urine of patients with rheumatoid arthritis and ankylosing spondylitis after single-dose intramuscular administration and its application to long-term pharmacokinetic study. J Pharm Biomed Anal. 2018 Feb 5;149:278-289. doi: 10.1016/j.jpba.2017.11.021. Epub 2017 Nov 6. PMID 29128828